CLINICAL TRIAL: NCT06487897
Title: Phase III Presbyopia Correction Using the VIS Optimal Keratoplasty (Opti-K™) System (Phase IIIa)
Brief Title: Phase III Presbyopia Correction Using the VIS Opti-K™ System
Acronym: Opti-K™
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: VIS, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OK-004
Record Dates: First submitted 2024-06-27; First posted 2024-07-05 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-08

CONDITIONS: Presbyopia
Keywords: Presbyopia,; Near Vision; Monovision; UNVA
MeSH Terms: conditions — Presbyopia; Myopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Single arm treatment with the VIS Optimal Keratoplasty (Opti-K™) System (Experimental): Subjects who accept monovision will receive Opti-K™ treatment in the non-dominant eye. The fellow eye will not receive Opti-K™ treatment in this Pivotal Study. Eligible subjects will undergo a single retreatment
  Interventions: Device: Optimal laser keratoplasty

INTERVENTIONS:
Device: Optimal laser keratoplasty — Laser

SUMMARY:
The goal of this clinical trial is to evaluate the safety and efficacy of using the VIS Opti-K System to enable monovision by providing temporary improvement in near vision through the treatment of the non-dominant eye of low myopic, emmetropic and low hyperopic presbyope subjects. The main questions it aims to answer are determining uncorrected near visual acuity at 40cm in the treated eye and subjective improvement as measured by the patient satisfaction questionnaire.

ELIGIBILITY:
Inclusion Criteria:

1. Subject age is equal to or greater than 40 years old.
2. Subjects must have a manifest refraction spherical equivalent (MRSE) between -0.5 D and +0.25 D with no more than 0.75 D of refractive cylinder needing +1.00 D to +2.50 D of reading add in both eyes.
3. Documented stable refractions defined as 0.5 D or less change in MRSE per year for 12 months or longer prior to primary Opti-K™ treatment, based on refractions, medical records, or prescription history.
4. Uncorrected distance visual acuity (UDVA) 20/25 or better (i.e., LogMAR ≤ 0.10) in both eyes.
5. Best corrected distance visual acuity (CDVA) of 20/20 or better (i.e., LogMAR ≤ 0.00) in both eyes.
6. Uncorrected near visual acuity (UNVA) between 20/50 (LogMAR 0.40) and better than 20/100 (LogMAR < 0.70) in the non-dominant eye.
7. Best corrected near visual acuity (CNVA) of at least 20/20 in both eyes (LogMAR ≤ 0.00).
8. Subject has normal corneal topography.
9. Subject must have documented monovision tolerance (per Appendix B)
10. Subject is not a contact lens wearer or, if wearing contact lenses, has discontinued wearing contact lenses for the required period of time and completed the contact lens stability check as described below.

    a. Contact Lens Wearers Only: Demonstration of a stable refraction, defined as two manifest refractions that are within ± 0.5 D MRSE of each other as determined under the following conditions: i. The two refractions are performed at least 7 days apart; and, ii. Contact lenses are not worn for at least the specified period prior to the first refraction used to establish stability and through the day of surgery:

    Contact Lens Type Minimum Discontinuation Time Soft 3 Days Soft Extended Wear 1 Week Soft Toric 2 Weeks Rigid gas permeable 2 Weeks
11. Subject is willing and able to comply with all pre-treatment and follow-up requirements, including the ability to read English to complete the PROWL questionnaire
12. Subject understands the nature of the procedure, as well as potential risks or limitations of the treatment, and provides informed consent.
13. Subject will make every effort to have no other refractive or ocular surgery during their study post-treatment follow-up period.

Exclusion Criteria:

1. Latent hyperopia 1.0 D (i.e., baseline MRSE and CRSE should not differ by or be more than 1.0 D or CRSE).
2. Nystagmus.
3. Significant conjunctivochalasis defined as laxity and/or looseness of the conjunctiva when traction is applied and/or redundancy in its normal state. If there is no redundancy of the conjunctiva under normal conditions, there should be no more than 3 mm of conjunctival movement on the bulbar surface in the cardinal fields of gaze and/or by displacement for the patient to qualify for enrollment.
4. Any active ocular surface disease of any severity.
5. Any condition causing a cloudy cornea (e.g., scarring, dystrophies, epithelial or stromal edema) or cloudy anterior chamber.
6. Allergy to anesthetics or post-treatment medications, including NSAIDS.
7. History or current evidence of chronic allergic reactions, tearing and/or ocular irritation that might confound the outcome or increase the risk of the study.
8. The use of systemic medications that may confound the outcome or increase the risk of the study, including, but not limited to corticosteroids, antimetabolites, amiodarone, chloroquine, isotretinoin, sumatriptan, or other medications that may affect healing.
9. Subjects with a recent history (within one week prior to treatment) of using topical ophthalmic medications containing preservatives (such as benzalkonium chloride, except for medications specifically required in this protocol) and/or other ocular drugs that are cytotoxic.
10. Those with ocular manifestations of acute or chronic illness that might increase the risk or confound the outcome of the study (e.g., diagnosed autoimmune disease, systemic connective tissue disease, clinically significant atopic disease, unstable diabetes mellitus and all diabetes with ocular involvement, etc.).
11. Pregnant, planning to become pregnant, or lactating women.
12. Subjects participating in other ophthalmic clinical trials during this clinical investigation.
13. Persons who, in the determination of the investigator, are not competent to understand the procedure or the actions asked of them as research subjects or have unrealistic expectations or are considered emotionally labile.
14. Persons who may not be able to complete the requirements of returning to the investigator's clinic over the period of the study, or who may be difficult to locate or contact on short notice. This does not preclude vacations or travel.
15. Subjects who are likely to be exposed to high levels of ultraviolet radiation (from sunlight, tanning lights, etc.) without protective eyewear during the one- year period following Opti-K™ treatment.
16. Presence or history of any other condition or finding that, in the opinion of the investigator, makes the subject unsuitable as a candidate for Opti-K™ treatment or study participation or may confound the outcome of the study.
17. Presence of a pupil irregularity (e.g., decentered pupil or irregular shape) in the eye to be treated that could predispose the eye to a centration error during the treatment.
18. Previous intraocular or corneal surgery of any kind in either eye, including any type of surgery for either refractive or therapeutic purposes.
19. Subjects using topical ophthalmic medications to treat presbyopia or plan to use these medications during the study follow-up period.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2024-09-30 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Uncorrected near visual acuity 2 or more lines or better | 3 months
  • The proportion of treated eyes (target: at least 50%) that achieve an uncorrected near visual acuity (UNVA) that is 2 or more lines better than Screening following treatment

SECONDARY OUTCOMES:
Binocular uncorrected near visual acuity | 3 months
  The proportion of eyes (target: at least 50%) that achieve a binocular uncorrected near visual acuity (UNVA) of 20/40 or better after the treatment

OTHER OUTCOMES:
Percentage of eyes that achieve UNVA | 3 months
  Percentage of eyes that achieve UNVA of 20/40 or better and 20/20 or better
Subjective improvement in vision | 3 months
  • Subjective improvement in visual experience as measured by subject satisfaction questionnaire related to near vision, distance vision, visual symptoms and overall satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Harry Glen, M.D., Study Director
Locations (4):
- United States (4):
  - Cohen Laser & Vision Center, Boca Raton, Florida
  - Claris Vision Eye Health, South Dartmouth, Massachusetts
  - The Cornea & Laser Eye Institute, Teaneck, New Jersey
  - OCLI Vision - Oceanside, Oceanside, New York

IPD SHARING:
Plan to Share IPD: Yes
There is a plan to make IPD and related data dictionaries available.
Supporting Information: Study Protocol
URL: https://www.viscorrect.com

REFERENCES:
- [Background] McDonald MB, Hersh PS, Manche EE, Maloney RK, Davidorf J, Sabry M; Conductive Keratoplasty United States Investigators Group. Conductive keratoplasty for the correction of low to moderate hyperopia: U.S. clinical trial 1-year results on 355 eyes. Ophthalmology. 2002 Nov;109(11):1978-89; discussion 1989-90. doi: 10.1016/s0161-6420(02)01255-1. PMID 12414402
- [Background] undefined
- [Background] Solomon KD, Fernandez de Castro LE, Sandoval HP, Biber JM, Groat B, Neff KD, Ying MS, French JW, Donnenfeld ED, Lindstrom RL; Joint LASIK Study Task Force. LASIK world literature review: quality of life and patient satisfaction. Ophthalmology. 2009 Apr;116(4):691-701. doi: 10.1016/j.ophtha.2008.12.037. PMID 19344821